CLINICAL TRIAL: NCT00006001
Title: Phase II Trial of SU5416 (NSC #696819) in Patients With Advanced Colorectal Cancer
Brief Title: SU5416 in Treating Patients With Metastatic or Locally Recurrent Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02345; UCCRC-NCI-52; NCI-52; CDR0000068009 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2004-05-26 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Semaxinib

ARMS (1):
- Arm I (Experimental): Patient receive SU5416 IV over 60 minutes twice weekly for 4 weeks. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: semaxanib

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
Phase II trial to study the effectiveness of SU5416 in treating patients who have metastatic or locally recurrent colorectal cancer. SU5416 may stop the growth of colorectal cancer by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective response rate and disease stabilization rates of patients with previously treated metastatic or locally recurrent colorectal cancer treated with SU5416.

II. Determine the median and overall survival and time to progression in this patient population receiving this treatment.

III. Determine the toxicity of SU5416 in these patients.

OUTLINE: This is a multicenter study.

Patient receive SU5416 IV over 60 minutes twice weekly for 4 weeks. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression.

Patients are followed every 2 weeks for 4 weeks.

PROJECTED ACCRUAL: A total of 17-37 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or locally recurrent adenocarcinoma of the colon or rectum
* Progressive disease as defined by new or progressive radiologic lesions
* Measurable disease at least 1 dimension as at least 20 mm with conventional techniques or at least 10 mm with spiral CT scan
* Lesions seen on colonoscopic examination or barium studies, bone metastases, CNS lesions, CEA levels and ascites are not considered measurable
* Lesion accessible for biopsy which is not within prior radiation port
* Known history of CNS metastasis allowed if patients have had treatment, are neurologically stable, and do not require oral or intravenous steroids or anticonvulsants, provided brain scan (CT or MRI) shows absence of active or residual disease
* If neurologic signs or symptoms suggestive of CNS metastasis, negative brain scan required

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: WHO 0-2
* Life expectancy: At least 12 weeks
* WBC at least 3,000/mm3
* Platelet count at least 75,000/mm3
* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance at least 60 mL/min
* No uncompensated coronary artery disease
* No history of myocardial infarction or severe/unstable angina within past 6 months
* No severe peripheral vascular disease associated with diabetes mellitus
* No deep venous or arterial thrombosis within past 3 months
* No pulmonary embolism within past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other significant uncontrolled underlying medical or psychiatric illness
* No serious active infections
* No concurrent second malignancy except for nonmelanoma skin cancer or carcinoma in situ of the cervix unless completed therapy and considered to be at less than 30% risk of relapse
* No history of severe allergic or anaphylactic reactions to paclitaxel or docetaxel

PRIOR CONCURRENT THERAPY:

* No more than 2 prior chemotherapy regimens for metastatic disease
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy
* No other concurrent investigational antineoplastic drugs
* No prior radiotherapy to only site of measurable disease
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* At least 30 days since other prior investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2000-08; Primary Completion 2007-02 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (10):
- United States (10):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Division of Hematology/Oncology, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana